CLINICAL TRIAL: NCT04842955
Title: Interventional Cross-over Study to Evaluate the Modulators of Efficacy of Alternating Current Brain Stimulation (tACS) in Patients With Alzheimer's Disease
Brief Title: Modulators of Gamma tACS in Alzheimer's Disease (Mod-GammAD)
Acronym: Mod-GammAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Barbara Borroni, Professor, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NP4479
Record Dates: First submitted 2021-03-10; First posted 2021-04-13 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's disease; transcranial Alternating Current Stimulation; Gamma stimulation; tACS
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real tACS (Experimental): Single session of gamma tACS (40 Hz) at 3 mA over the superior parietal cortex (Precuneus)
  Interventions: Device: Gamma tACS (40 Hz) over the superior parietal cortex
- sham tACS (Sham Comparator): Single session of sham tACS over the superior parietal cortex (Precuneus)
  Interventions: Device: Sham tACS over the superior parietal cortex

INTERVENTIONS:
Device: Gamma tACS (40 Hz) over the superior parietal cortex — Single session of gamma tACS (40 Hz) over the superior parietal cortex
  Arms: real tACS
Device: Sham tACS over the superior parietal cortex — Single session of sham tACS over the superior parietal cortex
  Arms: sham tACS

SUMMARY:
Brain oscillations are ubiquitous in the human brain and have been implicated in cognitive and behavioral states defined in precisely tuned neural networks. In neurodegenerative disorders, neurodegeneration is accompanied by changes in oscillatory activity leading to the emerging concept of neurological and psychiatric disorders as "oscillopathies". Alzheimer's disease, which accounts for the vast majority of age-related dementias, is characterised by a prominent disruption of oscillations in the gamma frequency band. The restoration of gamma oscillations by neural entrainment in animal models of Alzheimer's disease have shown a remarkable decrease in the pathological burden of amyloid and tau via increased microglial activity, resulting in a significant increase of cognitive performances.

Transcranial alternating current brain stimulation (tACS), is a neurophysiological method of non-invasive modulation of the excitability of the central nervous system that is having an increasingly numerous spectrum of potential therapeutic applications. Recent studies have demonstrated the effectiveness of this method in modulating the natural frequencies of cerebral oscillation, underlying multiple cognitive processes such as verbal memory, perception and working memory. On the basis of these premises, the treatment with gamma tACS is proposed in patients affected by Alzheimer's disease.

In this randomized, double-blind, sham-controlled, cross-over study, the investigators will evaluate the modulators of response on cognitive measure to a single stimulation with gamma tACS on the posterior parietal cortex in patients with Mild Cognitive Impairment due to Alzheimer's disease.

DETAILED DESCRIPTION:
Brain oscillations are ubiquitous in the human brain and have been implicated in cognitive and behavioral states defined in precisely tuned neural networks. In neurodegenerative disorders, neurodegeneration is accompanied by changes in oscillatory activity leading to the emerging concept of neurological and psychiatric disorders as "oscillopathies". Alzheimer's disease, which accounts for the vast majority of age-related dementias, is characterised by a prominent disruption of oscillations in the gamma frequency band. The restoration of gamma oscillations by neural entrainment in animal models of Alzheimer's disease have shown a remarkable decrease in the pathological burden of amyloid and tau via increased microglial activity, resulting in a significant increase of cognitive performances.

Transcranial alternating current brain stimulation (tACS), is a neurophysiological method of non-invasive modulation of the excitability of the central nervous system that is having an increasingly numerous spectrum of potential therapeutic applications. Recent studies have demonstrated the effectiveness of this method in modulating the natural frequencies of cerebral oscillation, underlying multiple cognitive processes such as verbal memory, perception and working memory.

On the basis of these premises, the treatment with gamma tACS is proposed in patients affected by Alzheimer's disease.

In this randomized, double-blind, sham-controlled, cross-over study, the investigators will evaluate the modulators of response on cognitive measure to a single stimulation with gamma tACS on the posterior parietal cortex in patients with Mild Cognitive Impairment due to Alzheimer's disease.

Subjects will be randomized in two groups, one receiving a single treatment with gamma tACS (40 Hz) first and the other receiving sham stimulation. After one week the treatments will be exchanged. Patients will be evaluated with neuropsychological tests and neurophysiological measures of cholinergic transmission. Modulators of response, including cognitive reserve, baseline impairment, apo-E genotype, MRI measures of atrophy and connectivity, electric field modelling, will be considered.

ELIGIBILITY:
Inclusion Criteria:

- Mild Cognitive Impairment due to Alzheimer's disease (according to Albert et al., Alzheimers Dement 2011).

Exclusion Criteria:

* Cerebrovascular disorders, previous stroke, hydrocephalus, and intra-cranial mass documented by MRI.
* History of traumatic brain injury or other neurological diseases.
* Serious medical illness other than AD
* History of seizures
* Pregnancy
* Metal implants in the head (except dental fillings)
* Electronic implants (i.e. pace-maker, implanted medical pump)
* Age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Changes in Rey Auditory Verbal Learning Test scores | Baseline (immediately before the intervention) - Immediately after the intervention
  Participants are given a list of 15 unrelated words repeated over five different trials and are asked to repeat. Another list of 15 unrelated words are given and the patient must again repeat the original list of 15 words and then again after 30 minutes.
  The score ranges from 0 (worse performance) to 15 (best performance).
Changes in Face-Name Associative Memory Test scores | During the intervention compared to sham comparator
  The Face-Name Associative Memory Test is a cross-modal associative memory test, it includes 20 face-name pairs. The administration procedure starts with the presentation of 20 faces with each name and participants should read the name underneath the faces and try to learn each face-name pair. After 5 minutes, the faces are shown one by one and participants are asked to recall the associated names from 4 different names. The correct number of pairs recalled is recorded.
  The score ranges from 0 (worse performance) to 20 (best performance).

SECONDARY OUTCOMES:
Change in SAI measurements | Baseline (immediately before the intervention) - Immediately after the intervention
  By using transcranial magnetic stimulation (TMS), the investigators will evaluate the effects of gamma tACS on short latency afferent inhibition (SAI), which is a marker of cholinergic transmission.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Borroni, MD, Principal Investigator — Azienda Ospedaliera Spedali Civili, Brescia; Alberto Benussi, MD, Principal Investigator — Azienda Ospedaliera Spedali Civili, Brescia
Locations (1):
- AO Spedali Civili, Brescia, BS, Italy

IPD SHARING:
Plan to Share IPD: Yes
All data, including outcome measure results, study protocol and statistical analysis plan, will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the study completion indefinitely.
Access Criteria: Reasonable request

REFERENCES:
- [Background] Fries P. Neuronal gamma-band synchronization as a fundamental process in cortical computation. Annu Rev Neurosci. 2009;32:209-24. doi: 10.1146/annurev.neuro.051508.135603. PMID 19400723
- [Background] Iaccarino HF, Singer AC, Martorell AJ, Rudenko A, Gao F, Gillingham TZ, Mathys H, Seo J, Kritskiy O, Abdurrob F, Adaikkan C, Canter RG, Rueda R, Brown EN, Boyden ES, Tsai LH. Gamma frequency entrainment attenuates amyloid load and modifies microglia. Nature. 2016 Dec 7;540(7632):230-235. doi: 10.1038/nature20587. PMID 27929004
- [Background] Adaikkan C, Middleton SJ, Marco A, Pao PC, Mathys H, Kim DN, Gao F, Young JZ, Suk HJ, Boyden ES, McHugh TJ, Tsai LH. Gamma Entrainment Binds Higher-Order Brain Regions and Offers Neuroprotection. Neuron. 2019 Jun 5;102(5):929-943.e8. doi: 10.1016/j.neuron.2019.04.011. Epub 2019 May 7. PMID 31076275
- [Background] Martorell AJ, Paulson AL, Suk HJ, Abdurrob F, Drummond GT, Guan W, Young JZ, Kim DN, Kritskiy O, Barker SJ, Mangena V, Prince SM, Brown EN, Chung K, Boyden ES, Singer AC, Tsai LH. Multi-sensory Gamma Stimulation Ameliorates Alzheimer's-Associated Pathology and Improves Cognition. Cell. 2019 Apr 4;177(2):256-271.e22. doi: 10.1016/j.cell.2019.02.014. Epub 2019 Mar 14. PMID 30879788
- [Background] Herrmann CS, Rach S, Neuling T, Struber D. Transcranial alternating current stimulation: a review of the underlying mechanisms and modulation of cognitive processes. Front Hum Neurosci. 2013 Jun 14;7:279. doi: 10.3389/fnhum.2013.00279. eCollection 2013. PMID 23785325
- [Derived] Benussi A, Cantoni V, Grassi M, Brechet L, Michel CM, Datta A, Thomas C, Gazzina S, Cotelli MS, Bianchi M, Premi E, Gadola Y, Cotelli M, Pengo M, Perrone F, Scolaro M, Archetti S, Solje E, Padovani A, Pascual-Leone A, Borroni B. Increasing Brain Gamma Activity Improves Episodic Memory and Restores Cholinergic Dysfunction in Alzheimer's Disease. Ann Neurol. 2022 Aug;92(2):322-334. doi: 10.1002/ana.26411. Epub 2022 Jun 6. PMID 35607946